CLINICAL TRIAL: NCT04869098
Title: Effects of an Evening PROtein PrEload on Blood Glucose, Metabolic Health, and Gut Hormone Release in Night ShIfT Workers (PROPENSITy)
Brief Title: Effects of an Evening PROtein PrEload on Metabolic Health in Night ShIfT Workers (PROPENSITy)
Acronym: PROPENSITy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, A/Prof Leonie Heilbronn, A/Prof, University of Adelaide
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: H-2020-131
Record Dates: First submitted 2021-04-26; First posted 2021-05-03 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes; Shift-work Disorder
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whey protein preload condition (Experimental): Participants will consume 30 g whey protein isolate powder (dissolved in water) 1-1.5 hr prior to their main evening meal every day for 12 days.
  Interventions: Dietary Supplement: whey protein
- Placebo condition (Placebo Comparator): Participants will consume an energy-matched mixed-nutrient placebo drink 1-1.5 hr prior to their main evening meal every day for 12 days,
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: whey protein — Protein drink containing 30g whey protein isolate powder (dissolved in water) consumed 1-1.5 hr prior to their main evening meal every day for 12 days, No other advice will be given.
  Arms: Whey protein preload condition
Dietary Supplement: Placebo — Energy-matched mixed-nutrient placebo drink consumed 1-1.5 hr prior to their main evening meal every day for 12 days. No other advice will be given.
  Arms: Placebo condition

SUMMARY:
This study will compare the effects of a whey protein supplement or a placebo consumed before the evening meal on health outcomes in night shift workers.

DETAILED DESCRIPTION:
Participants are assigned in random order to two conditions, for 12 days each. The interventions are 1) a 30g whey protein preload consumed 1-1.5 hr prior to their main evening meal every day for 12 days. No other advice will be given. 2) an identical mixed-nutrient drink matched for caloric content, taste and palatability consumed 1-1.5 hr prior to their main evening meal every day for 12 days(placebo). Conditions are separated by a 2-week washout period, during which participants will be encouraged to maintain their habitual diet and physical activity levels. Metabolic testing will be performed at baseline, and at the end of both conditions.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Night shift workers (with a minimum of 6 months in their current shift work schedule)
* 35-65 years
* BMI 28.0-35.0 kg/m2; waist circumference > 80cm
* Weight stable in the past 6 months

Exclusion Criteria:

* Those working standard day time hours only, or those who work less than three to four night shifts per fortnight on average
* Personal history and/or diagnosis of: diabetes, cancer, major psychiatric disorders, liver disease, gastro-intestinal surgery or disease (including malabsorption), eating disorders, anaemia, insomnia or cardiovascular disease, and/or any other condition deemed unstable by the study physician
* Taking medications known to alter body composition or metabolism, including (but not limited to): any medication used to lower blood glucose or antidiabetic medications (metformin, sulfonylureas, Glucagon-like peptide-1 (GLP-1) analogues [i.e. exenatide], thiazolidinediones or DPP-IV inhibitors [i.e. 'gliptins']), medications affecting weight, appetite or gut motility (i.e. diuretics, domperidone, cisapride, orlistat, phentermine, topiramate)
* Participants who are taking stable doses (i.e. > 12 months) of androgenic medications (i.e. testosterone) or SSRI's will not be excluded. Personal history/diagnosis (self-reported) of diabetes (type 1 or 2), major psychiatric disorders (schizophrenia, major depressive disorder, bipolar disorder, eating disorders), gastrointestinal disorders, haematological disorders (i.e. thalassemia, iron-deficiency anaemia) insomnia, or any other medical condition, deemed unstable by the study physician
* Pregnant, planning a pregnancy or breastfeeding
* Those who have lost or gained >5% of body weight in the last 6 months
* Those who consume four or more standard drinks on a single occasion at a 'daily or almost daily' occurrence
* current smokers of cigarettes/marijuana/e-cigarettes/vaporisers
* unable to comprehend the study protocol (i.e. due to English language or cognitive difficulties)

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Glycaemic response | 12 days (3 hours meal test)
  Change in glucose (AUC) following a standard breakfast

SECONDARY OUTCOMES:
24-hour glucose profiles | 12 days
  Change in 24-hour glucose profiles assessed by continuous glucose monitoring
Glucose variability | 12 days
  Change in 24-hour glucose variability (as SD, standard deviation) assessed by continuous glucose monitoring
Glucose variability | 12 days
  Change in 24-hour glucose variability (as CV, coefficients of variation) assessed by continuous glucose monitoring
Glucose variability | 12 days
  Change in 24-hour glucose variability (as MAGE, mean amplitude of gylcaemic excursions) assessed by continuous glucose monitoring
GLP-1 | 12 days (3 hours meal test)
  Change in GLP-1 (AUC) following a standard breakfast
GIP | 12 days (3 hours meal test)
  Change in GIP (AUC) following a standard breakfast
glucagon | 12 days (3 hours meal test)
  Change in glucagon (AUC) following a standard breakfast
Insulin | 12 days
  Change in fasting and postprandial insulin following a standard breakfast
Ghrelin | 12 days (3 hours meal test)
  Change in ghrelin (AUC) following a standard breakfast
PYY | 12 days
  Change in YY (AUC) following a standard breakfast
Adiponectin | 12 days
  Change in fasting adiponectin
C-Reactive Protein (CRP) | 12 days
  Change in fasting CRP
Blood lipids | 12 days
  Changes in blood lipid profile (total cholesterol, HDL-, LDL-cholesterol and triglycerides)
Blood pressure | 12 days
  Changes in systolic blood pressure and diastolic blood pressure
Resting metabolic rate | 12 days
  Changes in resting metabolic rate
respiratory quotient | 12 days
  Changes in respiratory quotient

CONTACTS AND LOCATIONS:
Overall Officials: Amy T Hutchison, PhD, Principal Investigator — University of Adelaide
Locations (1):
- University of Adelaide, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No